CLINICAL TRIAL: NCT05926726
Title: JWATM214，an Armored GPC3-directed CAR-T ，in the Treatment Amongst Subjects With Advanced Hepatocellular Carcinoma ：a Single-arm, Open-label，Dose-escalation Study
Brief Title: GPC3-directed CAR-T in the Treatment Amongst Subjects With Advanced Hepatocellular Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JWATM214001
Record Dates: First submitted 2023-04-04; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-05

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-GPC3 T cells (Experimental): The safety and efficacy of JWATM214 will be evaluated in a 'BOIN'-designed dose escalation approach. 3 CAR-T dose levels will be tested in this study: 1×10^8, 3×10^8, and 10×10^8, whereas the dosage 0.5×10^8 and 30×10^8 CAR-T cells will be selected as optional back-up doses for potential escalation or de-escalation.
  Interventions: Biological: CAR-GPC3 T cells

INTERVENTIONS:
Biological: CAR-GPC3 T cells — Subjects will undergo leukapheresis to isolate peripheral blood mononuclear cells (PBMCs) for the production of JWATM214 . During JWATM214 production, subjects will receive a preconditioning chemotherapy regimen of cyclophosphamide and fludarabine to deplete the lymphocytes. After lymphodepletion, subjects will receive single-dose treatment with JWATM214 by intravenous (IV) injection.

SUMMARY:
This is a single arm, open-label, dose escalation clinical study to evaluate the safety and efficacy of infused autologous armored GPC3-directed CAR-T in patients with advanced hepatocellular carcinoma refractory to prior systematic treatments.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years-old, male or female
2. Voluntarily willing to participate in the study and sign the written informed consent form
3. Life expectation ≥12 weeks
4. Eastern Cooperative Oncology Group (ECOG) performance status scale ≤1
5. Histologically-confirmed hepatocellular carcinoma (HCC)
6. No benefits from curative surgery or other local therapies are expected at screening, judged by investigators
7. Radiologically-confirmed progression disease after at least one prior line of systematic treatment and limited benefits from current guideline or consensus for hepatocellular carcinoma are expected at screening, judged by investigators
8. Fresh samples or FFPE, immunohistochemistry (IHC)-stained GPC-3 positive with intensity ++ or +++
9. Per RECIST v1.1, at least one measurable lesion
10. Manageable lung metastasis
11. Barcelona Clinic Liver Cancer (BCLC) stage C or B and Child-Pugh ≤7
12. No active HBV infections
13. Adequate organ functions
14. Adequate venous access for APH
15. Non-hematological AEs induced by previous treatment must have recovered to CTCAE ≤1, except for alopecia and peripheral neuropathy
16. Women of childbearing potential must agree to use an effective and reliable contraceptive method during 28 days prior to lymphodepletion to 1 year post infusion; Male patients who have not undergone vasectomy and have sexual activity with women of childbearing potential must agree to the use of a barrier contraceptive method since lymphodepletion to 1year post infusion, and sperm donation is prohibited during the study
17. Women of childbearing potential must have negative serum β-hCG test result at screening and 48 hours prior to lymphodepletion

Exclusion Criteria:

1. Cholangiocarcinoma or histological-mixed hepatocellular cholangiocarcinoma
2. Active brain metastasis
3. Primary lesion or infused lesions with the longest diameter ≥15cm, or other potential risk which might not be appropriate for further study treatment judged by the investigator
4. Another primary malignancy within 3 years (with some exceptions for completely-resected early-stage tumors)
5. Systematic autoimmune disorders requiring long-term systematic immunosuppression
6. Previously treated with any genetically engineered modified T cell therapy (TCR-T/CAR-T) or other CGT
7. Active HCV, HIV, or syphilis
8. History of organ transplant
9. Uncontrolled or active infection at screening, prior to APH, 72 hours prior to lymphodepletion or 5 days prior to JWATM214 infusion
10. With severe cardiovascular disease
11. History or presence of clinically-relevant CNS disorders
12. Current presence of hepatic encephalopathy
13. ≥G2 hemorrhage within 30 days prior to screening, or in need of long-term anticoagulants
14. Active digestive ulcer or gastrointestinal bleeding within 3 months prior to screening
15. Pregnant or lactating women
16. Not satisfying wash-out period for APH
17. Unable or unwilling to comply with the study protocol, judged by the investigator
18. Other situations implying that the subject might not be appropriate to participate in the study
19. Previously allergic or intolerable to JWATM214 or its components

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment-related adverse events (AEs) | 2 years
  An AE is defined as any unfavorable and unintended sign, symptom, or disease (new or worsening) temporally associated with the use of study therapy, regardless of whether or not a causal relationship with the study therapy can be determined.
Dose-limiting toxicities | 28 days
  DLT (Dose-limiting toxicity) was an adverse event that occurred within 28 days after JWATM214 infusion that met any of the following criteria.
  1. Any grade ≥3 nonhematologic toxicity associated with JWATM214 that has not resolved to ≤ grade 2 within 7 days, excluding clinically insignificant abnormalities in laboratory indicators
  2. Hematologic toxicity
  3. Grade ≥3 anaphylaxis
  4. Grade ≥3 infection did not resolve to grade ≤2 within 7 days after anti-infective treatment.
  5. ≥ grade 3 autoimmune toxicity during treatment
  6. Grade ≥3 cytokine release syndrome (CRS) during treatment that did not resolve to grade ≤2 within 72 hours.
  7. Grade ≥3 CAR-T cell-associated encephalopathy syndrome/immune effector cell-associated neurotoxicity syndrome (CRES/ICANS) that did not resolve to grade ≤2 within 72 hours.
  8. Grade 5 events of any nonmalignant cause.
RP2D of JWATM214 in HCC patients | 2 years
  Recommended phase 2 dose of JWATM214

SECONDARY OUTCOMES:
PK of JWATM214 in the peripheral blood (qPCR) | 1 years
  The pharmacokinetic parameters of JWATM214 will be evaluated by qPCR for the copy number of the vector transgene of JWATM214 in peripheral blood to evaluate T-cell expansion and persistence.
Objective response rate (ORR). | 1 years
  Proportion of patients whose tumor volume has reached a predetermined value and can maintain a minimum time limit, including complete response and partial response patients.
Disease Control Rate | 2 years
  the percentage of patients with advanced or metastatic cancer who have achieved complete response, partial response and stable disease to a therapeutic intervention in clinical trials of anticancer agents.
progression-free survival (PFS) | 2 years
  Defined as time from randomisation to first progression by investigator assessment using modified RECIST 1.1 or death (by any cause in the absence of progression)
overall survival (OS) | 2 years
  Defined as the time from randomisation to death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Xia, Prof. MD, Study Chair — Dept. Liver Surgery, Renji Hospital, School of Medicine, SJTU; Hao Feng, MD.,Ph.D., Principal Investigator — Dept. Liver Surgery, Renji Hospital, School of Medicine, SJTU
Locations (1):
- Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided